CLINICAL TRIAL: NCT05684016
Title: Assessment of Deep Gray Matter Anatomic Changes in Relapsing Remitting Multiple Sclerosis (RRMS) Patients Treated With Gilenya® (Fingolimod) With and Without Cognitive Impairment Over a 2 Year Period Using 3 Dimensional Volumetric MRI Studies (NeuroQuant, NeuroQuarc) and Automated Neuropsychological Assessment Matrices (ANAM)
Brief Title: Assessment of Deep Gray Matter Anatomic Changes in RRMS Patients Treated With Gilenya® With and Without Cognitive Impairment Over a 2 Year Period Using NeuroQuant, NeuroQuarc and ANAM
Acronym: NeuroQuant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Ted Rothstein, Associate Professor of Neurology, George Washington University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ADEG-MS-3DV
Record Dates: First submitted 2015-01-08; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Relapsing Remitting Multiple Sclerosis; RRMS; Gilenya; Fingolimod; MRI; NeuroQuant; NeuroQuarc; Automated Neuropsychological Assessment Matrices; ANAM
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): A control population (Non RRMS) will include a minimum of 20 age and gender matched healthy patients from the George Washington University (GWU) neurology outpatient clinic (being compared with those RRMS patients being treated with Gilenya® ) for whom Brain MRI's are being ordered as a result of their having headaches, dizziness, or other conditions where there is no physical evidence for neurologic impairment. All control patients will only be recruited by the full time Neurology Faculty at the GWU Medical Faculty Associates (MFA). Control patients will be asked to consent to have NeuroQuant added to their routine Brain MRI which will add 7 minutes to their time in the MRI scanner to obtain additional image data.
  Interventions: Other: NeuroQuant; Other: Automated Neuropsychological Assessment Matrices
- MS Subject on Gilenya (Active Comparator): All the RRMS patients will have their Brain MRI with the addition of NeuroQuant. The 30 patients that are taking Gilenya® will have serial NeuroQuant/MRI and Neuropsychological testing (which is like an IQ test) using Automated Neuropsychological Assessment Matrices (ANAM) whether they are or are not experiencing cognitive issues. In addition, each study patient will undergo Extended Disability Status Score (EDSS) evaluation by a physician or a physician assistant at baseline and at 1 and 2 years. A group of 20 RRMS patients will undergo a second Brain MRI (not standard of care) with NeuroQuant evaluation 7 to 14 days after the initial study in order to confirm the reproducibility of this imaging technique. The cost for this repeat MRI will not be charged to you but will be borne by the sponsors of this study
  Interventions: Other: NeuroQuant; Other: Automated Neuropsychological Assessment Matrices; Other: EDSS; Other: Physical Examination
- MS Subject not on Gilenya (Active Comparator): All the RRMS patients will have their Brain MRI with the addition of NeuroQuant.
  Interventions: Other: NeuroQuant; Other: EDSS; Other: Physical Examination

INTERVENTIONS:
Other: NeuroQuant — Reliably defines the volume of those parts of the brain that are important for memory and thinking.
Other: Automated Neuropsychological Assessment Matrices — This is like an IQ test.
  Arms: Control; MS Subject on Gilenya
Other: EDSS — Extended Disability Status Score
  Arms: MS Subject not on Gilenya; MS Subject on Gilenya
Other: Physical Examination — Physical Examination
  Arms: MS Subject not on Gilenya; MS Subject on Gilenya

SUMMARY:
The purpose of the research study is to investigate whether the extent and severity of lesions in the brain as measured by special MRI techniques can distinguish between Multiple Sclerosis (MS) patients with or without memory impairment and also between MS patients and age matched healthy controls.

DETAILED DESCRIPTION:
Impairment in thinking or memory is frequently present in multiple sclerosis but there are difficulties finding changes on the Brain MRI that correlate with impairment in thinking and memory. This occurs because standard MRI is good for detecting some but not all abnormalities in the brain. Those lesions that we do see in the brain on standard MRI do not correlate with memory impairment or the source of disability in most RRMS patients. This occurs because RRMS symptoms mainly result from parts of the brain which have been hard to evaluate with MRI until now.

To gain more insight into the source of memory impairment, we plan to explore differences in brain volume that may be present in RRMS patients without thinking or memory problems compared with those who are impaired. A secondary objective will be to compare RRMS patients in general with healthy controls.

A new MRI technique called NeuroQuant which reliably defines the volume of those parts of the brain that are important for memory and thinking will be used. Neuropsychological testing will also be offered, at no cost, to those patients being treated with Gilenya® in order to help define the presence and extent of their memory impairment. Automated Neuropsychological Assessment Matrices (ANAM)looks at all functional brain systems and will be administered by a psychometrist over a period of 90 minutes.

ELIGIBILITY:
Inclusion and Exclusion Criteria

RRMS Patients

Inclusion Criteria

* Male and Female adult definite RRMS patients with or without cognitive complaint
* Age range 18-55 years old
* Patients treated with Gilenya® (fingolimod) and other immunomodulating MS therapies
* Able to provide informed consent

Exclusion Criteria

* Pregnant or breastfeeding women
* Patients with an infectious disease
* Patients with any other medical or neurological condition that could affect cognition
* Inability to communicate in English
* Patients with clinically or radiologically isolated syndrome (CIS, RIS)
* Primary or Secondary Progressive forms of MS
* Current or past medical, neurological or psychiatric disorders (other than MS)
* Previous illicit substance dependence or substance abuse
* Pulse or steroid therapy within 8 weeks or preceding evaluation
* Current major depressive episode

Control Patients

Inclusion Criteria

* Male and Female adult with normal brain MRI and Neurological Examination
* Headaches or dizziness
* Age range 18-55 years
* Able to provide informed consent

Exclusion Criteria

* Patients with an infectious disease
* Patients with any other medical or neurological condition that could affect cognition
* Inability to provide informed consent
* Inability to communicate in English
* Pregnant or breastfeeding woman

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2013-12; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Changes in size of brain region by cm3 over a 2 year period in RRMS patients with and without cognitive impairment compared to healthy age matched controls | 2 Years
  a. Utilizing MRI 3 dimensional volumetric analysis (NeuroQuant) to detect gray matter changes in RRMS with or without cognitive impairment and compare results with normal demographically similar age matched controls.

SECONDARY OUTCOMES:
Determine in patients with RRMS treated with Gilenya®, the changes on various gray matter volume as assessed by serial NeuroQuant/NeuroQuarc 3 dimensional volumetric analysis over a 2 year period. | 2 Years
  a. Use serial MRI 3 dimensional volumetric analysis (NeuroQuant) at baseline, 1 week (in 20 patients) and 1 and 2 years to assess reproducibility of NeuroQuant, and determine the degree of preservation of gray matter structures in RRMS patients treated with Gilenya® over a period of 2 years.
Compare Neuropsychological Evaluations using ANAM to address cognitive changes in patients treated with Gilenya over time as compared to healthy aged matched control patients. | 2 years
  Baseline neuropsychological evaluations on patients treated with Gilenya based on results of an Automated Neuropsychological Assessment Matrices (ANAM). Healthy controls will also undergo this neuropsychological assessment. Both groups will be repeatedly tested over time for 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Ted Rothstein, MD, Principal Investigator — The George Washington University
Locations (1):
- The George Washignton University, Washington D.C., District of Columbia, United States